CLINICAL TRIAL: NCT05436483
Title: Preliminary Establishment of the Medical Reference Range of Serum Vitamin K2 in Chinese Healthy Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022008
Record Dates: First submitted 2022-06-20; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-04

CONDITIONS: Health, Subjective

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteocalcin is a type of vitamin K2-dependent protein, and many studies have confirmed that vitamin K2 has anti-osteoporosis effects, and has preventive and therapeutic effects on a variety of diseases such as nervous system, cardiovascular disease, immune disease, and glucose metabolism. However, as a pleiotropic vitamin and nutrient, vitamin K2 does not have an exact normal range like other vitamins, when it needs to be supplemented, and in what regimen. Different organizations have different opinions on the recommended intake of vitamin K. Thus, this study intends to preliminarily obtain the reference interval of serum vitamin K2 by conducting clinical research in healthy people in the Beijing-Tianjin-Hebei region, and analyzes different factors, such as gender, age, and place of residence, to compare their level differences and changing trends, and to provide data reference for the recommended intake of vitamin K2 for people with vitamin K2 deficiency.

ELIGIBILITY:
Inclusion Criteria:

* People aged over 18.
* People with normal routine blood test.
* Willing to participate in this study.

Exclusion Criteria:

* Subjects with congenital metabolic problems and endocrine diseases.
* Treatment with any investigational drug within the past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 465 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of vitamin K2 | During the procedure of regular physical checkups
  Vitamin K2 concentration in serum